CLINICAL TRIAL: NCT00718367
Title: Correlation of the Clinical Behaviour of Renal Cell Carcinoma (RCC) After Debulking Nephrectomy With Tumor Gene Expression in Nephrectomy Specimens
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: RC01/31/07
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The objective of the study is to determine whether a specific immune microenvironment in the primary tumor is associated with a favorable clinical course after nephrectomy and in the absence of adjuvant treatment.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is a tumor with clinically apparent immunologic phenomena, such as response to immunotherapies (interferon, interleukin-2, immune cellular therapy etc), spontaneous regression, and sometimes indolent behaviour. Nephrectomy itself influences the prognosis of advanced RCC patients as shown in 2 randomised trials, and could have an immune basis. We previously reported on the variability of clinical behaviour in advanced RCC patients who had not received systemic treatment after debulking nephrectomy (Debulking Nephrectomy Followed By A "Watch And Wait" Approach In Metastatic Renal Cell Carcinoma .Wong A, et al. Urol Oncol, in press). The clinical significance of this includes the avoidance of toxic systemic therapies after nephrectomy, or the possibility of using non-toxic vaccine approaches in metastatic patients after cytoreductive nephrectomy. In this research proposal we would like to analyse the immune related gene expression profile on nephrectomy tumor samples and correlate them with the clinical course of the patient after the nephrectomy. This will be an exploratory and retrospective study of 15 patients in whom debulking nephrectomy for advanced RCC had been done, who did not receive any adjuvant treatment, and in whom the clinical course had been monitored after the nephrectomy.

We will first carry out a feasibility study during which we will isolate RNA from 3 FFPE (formalin-fixed,paraffin-embedded) samples using commercially available RNA isolation kit and we will determine if their quality is compatible with quantitative polymerase chain reaction (qPCR) or microarray studies. Upon successful feasibility study, the analysis will be extended to 15 patients. RNA will be isolated from FFPE samples and the gene expression profiles will be evaluated by qPCR and/or microarray. Emphasis will be placed on the expression profile of immune-related genes. Finally, transcriptome analysis results will be extended at the protein and cell level using immunohistochemistry assays.

ELIGIBILITY:
Inclusion Criteria:

* Advanced RCC who had a cytoreductive nephrectomy done.
* Patients did not receive specific anti-cancer systemic therapy after the nephrectomy, except after clinical disease progression.
* Tumor samples available.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced RCC who had a cytoreductive nephrectomy done. Patients did not receive specific anti-cancer systemic therapy after the nephrectomy, except after clinical disease progression. Tumor samples available.
Sampling Method: Non-Probability Sample
Dates: Start 2008-03; Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Seng Cheong Wong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore; Sing Joo Chia, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Kondo T, Nakazawa H, Ito F, Hashimoto Y, Osaka Y, Futatsuyama K, Toma H, Tanabe K. Favorable prognosis of renal cell carcinoma with increased expression of chemokines associated with a Th1-type immune response. Cancer Sci. 2006 Aug;97(8):780-6. doi: 10.1111/j.1349-7006.2006.00231.x. PMID 16863511